CLINICAL TRIAL: NCT05310422
Title: Safety Study of Tivanisiran to Treat Dry Eye
Acronym: FYDES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYL1001_VI
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Disease
Keywords: siRNA; oligonucleotide; keratoconjunctivitis sicca; SYL1001
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tivanisiran sodium ophthalmic solution (Experimental)
  Interventions: Drug: Tivanisiran sodium ophthalmic solution
- Vehicle ophthalmic solution (Placebo Comparator)
  Interventions: Drug: Vehicle ophthalmic solution

INTERVENTIONS:
Drug: Tivanisiran sodium ophthalmic solution — 1 drop in the affected eye(s) once daily
  Arms: Tivanisiran sodium ophthalmic solution
Drug: Vehicle ophthalmic solution — 1 drop in the affected eye(s) once daily
  Arms: Vehicle ophthalmic solution

SUMMARY:
This study will examine the safety of tivanisiran sodium eye drops versus vehicle when dosed once daily for 1 year in subjects with signs and symptoms of dry eye disease (DED).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have given their written consent to participate in the study
* Use of artificial tears (AT), autologous serum or specific dry eye medications during the last 6 months prior to the selection

Exclusion Criteria:

* Pregnant or breast feeding females with a postitive pregnancy test
* Women of childbearing potential not willing to use a medically acceptable contraceptive method
* Currently participating or has participated in another clinical trial within the 2 months prior to inclusion
* Current, previous chronic or recurrent medical condition that, according to the investigator, might impact on the study
* Any concomitant treatment or prior ocular procedure or surgery in either eye or alteration of the dose of systemic medications that could interfere in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Frequency and percentage of subjects with ocular and non-ocular treatment emergent adverse events (TEAEs) for 1 year | 1 year

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Sylentis Investigative Site, Chandler, Arizona
  - Sylentis Investigative Site, Phoenix, Arizona
  - FYDES Investigative Site, Glendale, California
  - Sylentis Investigative Site, Hemet, California
  - Sylentis Investigative Site, Los Angeles, California
  - Sylentis Investigative Site, Murrieta, California
  - Sylentis Investigative Site, Newport Beach, California
  - FYDES Investigative Site, Delray Beach, Florida
  - FYDES Investigative Site, Jacksonville, Florida
  - Sylentis Investigative Site, Largo, Florida
  - Sylentis Investigative Site, Morrow, Georgia
  - Sylentis Investigative Site, Fraser, Michigan
  - Sylentis Investigative Site, Kansas City, Missouri
  - FYDES Investigative Site, St Louis, Missouri
  - Sylentis Investigative Site, Washington, Missouri
  - Sylentis Investigative Site, Rochester, New York
  - Sylentis Investigative Site, Asheville, North Carolina
  - Sylentis Investigative Site, Garner, North Carolina
  - Sylentis Investigative Site, Cranberry Township, Pennsylvania
  - Sylentis Investigative Site, Rapid City, South Dakota
  - Sylentis Investigative Site, Memphis, Tennessee
  - Sylentis Investigative Site, Austin, Texas
  - FYDES Investigative Site, El Paso, Texas
  - Sylentis Investigative Site, San Antonio, Texas

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473